CLINICAL TRIAL: NCT02790827
Title: Randomized Controlled Trial of a Multi-pronged Intervention to Address Prevention of Violence in Zambia
Brief Title: Trial of a Multi-pronged Intervention to Address Prevention of Violence in Zambia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: SHARPZ (Serenity Harm Reduction Programme Zambia) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00006534
Record Dates: First submitted 2016-05-24; First posted 2016-06-06 (Estimated); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Domestic Violence; Mental Health Impairment; Child Abuse; Alcoholism
MeSH Terms: conditions — Alcoholism | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CETA (Experimental): Participants in the experimental arm will receive the CETA intervention. The intervention period will last for approximately 4 months with weekly sessions. There will be separate groups for men, women, and children. Each group will have approximately six participants. Individuals who cannot attend group therapy (e.g., conflicting work schedules) may be offered the therapy individually.
  Interventions: Behavioral: CETA
- Treatment as usual (Active Comparator): There is no standard of care for domestic violence or alcohol use problems in Zambia. We will track any treatment or care that families receive during the course of the study. The active comparator arm will not receive any formal services provided by the study.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: CETA — CETA first focuses on: 1) awareness of alcohol problems, violence, and the link between them; 2) gender norms. Skills taught include: changing drinking behaviors, coping with cravings, family dynamics that contribute and result from alcohol use, the role gender plays, and community norms around problem drinking, and cognitive/emotional/behavioral patterns connected with inter-personal violence. The intervention then addresses: 1) positive parenting, 2) positive family relationships, conflict management, and communication skills, 3) attitudes and beliefs about violence, 4) mental health problems and 5) reducing (further) traumatic experiences. The cognitive behavioral therapy (CBT) principles of CETA overlap with the CBT skills for alcohol reduction.
  Arms: CETA
Behavioral: Treatment as usual — The control condition is defined as 'treatment as usual'. In Zambia, there are no formal services or standard of care for alcohol use problems or domestic violence. There are, however, organizations (such as non-governmental organizations) operating in Lusaka that provide intermittent services for these types of problems. Some families receive informal counseling from parish priests or other leaders in their communities. In this study we are therefore defining these types of informal services as 'treatment-as-usual.' We will closely track the type, number, and degree of these kinds of services that all participants receive and access. Following the conclusion of the study, we will offer the CETA intervention to control families if it has been found to be safe and effective.
  Arms: Treatment as usual

SUMMARY:
This study evaluates the effectiveness of a multi-pronged intervention in reducing and preventing violence against women and children compared to a treatment as usual control group among families living in Lusaka, Zambia.

DETAILED DESCRIPTION:
Aims:

1. To test the effectiveness of a multi-pronged intervention in reducing and preventing violence against women and children compared to a treatment as usual control group among families living in Lusaka, Zambia.
2. To test the effectiveness of a multi-pronged intervention compared to a treatment as usual control group in reducing identified risk factors of violence including alcohol use, mental health problems, poor parenting skills, and family communication and behavior patterns.

Design Overview:

This is a randomized controlled trial to evaluate the effectiveness of a multipronged intervention in reducing violence against women and girls/youth (VAWG) by addressing a number of identified risk factors (e.g., childhood abuse, domestic violence, alcohol use). 168 families from compounds (i.e. communities) in the city of Lusaka will be randomized to either control or experimental condition. An adult male, adult female, and one child from each family will be a "unit" and participate in the study. Child participation is optional (i.e., the adult male and female in the family unit may participate if they don't have children or do not provide permission for a child to participate).

The experimental intervention, a cognitive behavioral therapy-based psychotherapy (CETA) focuses on alcohol abuse and gender-specific violence, and addresses mental health, abuse, parenting skills, family communication and behavior patterns. There may be conjoint sessions that include both caregiver(s) and child(ren), when and if possible. During the 4-5 month intervention period there will be three group sessions per week: one for a male group, one group for women, and one group for children. Each counseling group will have approximately six group members. The intervention is designed this way due to research supporting multi-modal treatments, and to model how organizations are likely to incorporate a program to prevent violence into its regular services (i.e., group-based vs. individual sessions). The primary outcomes of the study are severity of violence against women and children. Secondary outcomes include alcohol use aggression, mental and behavioral health and gender norms.

The control condition is defined as 'treatment as usual'. In Zambia, there are no formal services or standard of care for alcohol use problems or domestic violence. There are, however, organizations (such as non-governmental organizations) operating in Lusaka that provide intermittent services for these types of problems. Some families receive informal counseling from parish priests or other leaders in the communities. In this study investigators are therefore defining these types of informal services as 'treatment-as-usual.' Investigators will closely track the type, number, and degree of these kinds of services that all participants receive and access. Following the conclusion of the study, investigators will offer the CETA intervention to control families if it has been found to be safe and effective.

Participants:

Participants will be family units consisting of three individuals: an adult woman, her husband or partner, and one identified child if the adult couple chooses to include a child in the study (children may be male or female, ages 8-17, and should be described by the adult female as the child most affected by violence). The families will be recruited from urban communities (compounds) in Lusaka where violence and alcohol abuse are known to be problems. A family will be included in the study if the adult female indicates in a brief screener a moderate amount of violence within the family as measured by scoring a 38 or more on the Severity of Violence Against Women Scale (SVAWS). The male in the family must also indicate that he drinks alcohol at hazardous levels and/or the female must indicate that the male drinks alcohol at hazardous levels as evidenced by a score of 8 or higher on the Alcohol Use Disorders Identification Test (AUDIT). The man and the woman must agree to participate in the study in order for the family to be eligible. The participation of the child is optional. The parents may decide to participate but not provide permission for the parents' child to participate. The child may also choose not to participate him/herself. In either case, the parents may still be included in the study without the child.

Recruitment:

Study participants will be recruited from urban communities through several methods.

The primary method of recruitment will be outreach by CETA counselors. The CETA counselors who are recruited and trained by Johns Hopkins University (JHU) and Serenity Harm Reduction Programme Zambia (SHARPZ) to conduct the interventions have deep ties within the communities and have knowledge of families that may benefit from the intervention. The CETA facilitator will go door-to-door and approach families in the community that s/he thinks can benefit from the intervention. This is the current standard procedure for the similar programs run through SHARPZ in other Lusaka communities. The counselor will ask the family if there is a time the family could meet privately to discuss the study and the CETA services. The meeting will take place at a time and place that is convenient for the family. Investigators will provide the CETA facilitators with a recruitment script to give an overview of the study and CETA intervention to the family.

Investigators will also include three other recruitment strategies as necessary.

One of these additional strategies will be through church-based and community leader outreach efforts in the compounds. In Lusaka, community leaders in the compounds are often associated with the local churches. Investigators will hold community meetings in which investigators describe the study and its purpose in general terms to community members. Investigators will then advertise a designated time and place (typically at the local parish) where interested families can come and speak to research staff about participating in the study and to receive full information about participation. Investigators will also ask Home Based Care Workers (HBCWs) working with these churches to discuss the study with families for whom they already provide care. Investigators will ask the HBCWs to do this using the same recruitment script as the CETA counselors. Families who are interested in hearing more about the study after speaking with the HBCW will be able to meet research staff at the designated place/time for full study information, consent, and screening procedures. Recruitment through churches and with HBCWs has been effective in previous studies investigators have conducted in Zambia and has been found to be acceptable by the communities in Lusaka.

A second additional strategy will be through a snowball sampling method. Investigators may ask participants who have been enrolled into the study to refer other families, neighbors, and community members who may be affected by violence or alcohol abuse to us. Investigators will provide the current participants with information on the next designated place and time of study assessments and can pass this information off to others in the community. Investigators will also provide contact information in case potential participants want to contact us directly. Investigators have found in previous studies in Zambia that participants often come to us to ask if participants may refer other friends or neighbors to the study for participation.

A third strategy may include referral by on-going community support groups in the compounds. Members of these groups often have information about families in the communities who may have problems with violence and/or alcohol. Investigators will provide information to these groups about the next day/time assessments will be conducted in the area and ask them to pass on that information to other families.

In all of the above strategies, potential study participants will have no contact with research study staff until participants express to someone (i.e., the CETA counselor, a HBCW, or a friend/neighbor who is already enrolled) interest in hearing more about the study and would like the research staff to contact them.

If the family is eligible for the study, each member will be assigned a unique study identification (ID) number. These ID numbers will be used to start the ACASI (laptop-based) assessment for each participant. Participants will complete the assessments separately and privately using the ACASI laptops and with headphones.

No identifying information (names, addresses, phone numbers) will be captured by ACASI. Following the completed assessment, the three ID numbers will be brought to the SHARPZ main office by the study assessor, where ID numbers will be securely stored by the Study Director. The Study Director will forward eligible ID numbers each day to JHU-based research staff who will randomly allocate each family (cluster of 3 ID numbers) to either intervention or control condition. The family will be notified by the study team within one day following the baseline assessment of the randomization assignment. If participants are assigned to the control group, investigators will explain procedures for calling them weekly to check in for the next several months (during the active intervention phase) and monthly thereafter for the next two years while the study is on-going. If participants were randomized to the intervention, Investigators will let participants know that investigators will be contacting them within a week and weekly thereafter with details about starting the group counseling sessions (groups are expected to begin within approximately 3 weeks following assessment).

Assessments of violence, alcohol use, and other secondary outcomes will be conducted at four timepoints using ACASI:

1. Baseline
2. 4-5 months post-baseline (immediately following intervention period)
3. 12 months post-baseline
4. 24 months post-baseline (primary timepoint of interest)

Descriptions of self-report outcome measures are described below. In addition to the self-report measures captured through ACASI, investigators will collect a hair-sample from each participant at all four time points to test for cortisol, a well-established biomarker for chronic stress.

The primary timepoint of interest is the 24 month assessment. The Data and Safety Monitoring Board (DSMB) will will conduct an analysis at the 12 month assessment to assess effectiveness of CETA in reducing violence. If there is a statistically and clinically significant effect, the trial will be stopped and investigators will offer the intervention to the control participants. Investigators would then assess outcomes at the 24 month assessment among intervention participants to monitor whether treatment effects were sustained.

Sample size calculations are based on the SVAWS measure. Calculations are based on a recent study conducted in South Africa with women who had been abused by a partner who had an alcohol use problem. The study found a mean SVAWS physical violence sub-scale score of 58.6 (SD=20.5) with a time reference of the past three months. Investigators believe that a 20% reduction in the mean SVAWS physical violence subscale score would be programmatically significant (i.e. worth finding). The sample size needed to obtain an 11.66 point reduction among intervention participants at 12 months, assuming no change among control participants, with 80% power and an alpha of 0.05, is 100 families (50 per arm). To account for potential drop-out/loss to follow-up and potentially small clustering effects at the provider/group level, investigators aim to recruit 84 families in each trial arm, for a total of 168 families enrolled in the study.

All analyses will be intent to treat. For each continuous outcome (e.g., SVAWS score) investigators will estimate linear mixed effects models that will incorporate a random intercept term to account for within subject correlation on repeated measures. Generalized linear models will be used for categorical outcomes. The outcome scores at the follow-up times will be modeled separately using treatment arm, baseline symptom score (if there is a meaningful difference between the study arms at baseline), time, and an interaction between each treatment arm and time as fixed covariates in each model.

Protocol update October 2016:

Following the first few weeks of intervention delivery, investigators found that for a significant number of participants, group therapy sessions were impractical due to logistical challenges. Therefore, investigators modified the delivery of CETA for some participants to be individually delivered therapy sessions instead of group therapy sessions. Participants who are able to attend group sessions and prefer that method will still receive the intervention through the group delivery method.

The sample size was increased in order to have statistical power to conduct a sub-group analysis of only those study participants who received individual (and not group) CETA to test whether this individual delivery mode is effective compared to the treatment as usual control group. An additional 80 families (40 randomized to each arm) will be recruited into the study for this purpose. The total sample size is therefore planned to be 248 families.

ELIGIBILITY:
Inclusion Criteria:

1. Families living in the study compounds in Lusaka (i.e., not staying temporarily)
2. Speaking one of the three study languages: English, Bemba, or Nyanja
3. Having at least one male adult and one female adult 18 years of age or older and in a relationship (married or dating) and one child between the ages of 8 to 17 identified by the mother as the most affected by the violence (if multiple children in the home). Child participation is optional.
4. The man and woman must both provide consent. If the female agree to have the child participate and the child wants to participate, then parental permission and child assent will be required.
5. The adult female must indicate during the inclusion screening at least a moderate amount of violence within the family as measured by scoring a 38 or more on the Severity of Violence Against Women Scale (SVAWS).
6. The male in the family must indicate that he drinks alcohol at hazardous levels or the female must report that the male drinks alcohol at hazardous levels as evidenced by scoring an 8 or higher on the Alcohol Use Disorders Identification Test (AUDIT).

Exclusion Criteria:

1. Any of the family members is currently on an unstable psychiatric drug regimen (i.e., regimen altered in last 2 months)
2. Any of the family members has had a suicide attempt or suicidal ideation with intent or plan, or self-harm in the past month.
3. Any of the family members has been diagnosed with a current psychotic disorder (identified by the University Teaching Hospital Psychiatric Unit).
4. Any of the family members has a serious developmental disorder (e.g., mental retardation, autism) that would preclude participation in cognitive-behavioral oriented skills intervention

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 626 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Change in violence against women as measured by Severity of Violence Against Women Scale (SVAWS) | Baseline, 4-5 months post-baseline, 12 months post-baseline, 24 months post-baseline

SECONDARY OUTCOMES:
Change in alcohol abuse as measured by the Alcohol Use Disorders Identification Test (AUDIT) | Baseline, 4-5 months post-baseline, 12 months post-baseline, 24 months post-baseline
Change in child abuse as measured by the Youth Victimization Scale | Baseline, 4-5 months post-baseline, 12 months post-baseline, 24 months post-baseline
Change in depression symptoms as measured by the Center for Epidemiological Studies Depression Scale (CES-D) | Baseline, 4-5 months post-baseline, 12 months post-baseline, 24 months post-baseline
Change in PTSD symptoms (adult) as measured by the Harvard Trauma Questionnaire (HTQ) | Baseline, 4-5 months post-baseline, 12 months post-baseline, 24 months post-baseline
Change in belief about gender norms as measured by the Gender Equitable Mens Scale (GEMS) | Baseline, 4-5 months post-baseline, 12 months post-baseline, 24 months post-baseline
Change in child internalizing and externalizing symptoms as measured by the Youth Self Report (YSR) | Baseline, 4-5 months post-baseline, 12 months post-baseline, 24 months post-baseline
Change in substance use as measured by the Alcohol, Smoking, and Substance Involvement Screening Test (ASSIST) | Baseline, 4-5 months post-baseline, 12 months post-baseline, 24 months post-baseline
Change in child aggression as measured by the Child Aggression Scale | Baseline, 4-5 months post-baseline, 12 months post-baseline, 24 months post-baseline
Change in PTSD symptoms (child) as measured by the Child PTSD Symptom Scale (CPSS) | Baseline, 4-5 months post-baseline, 12 months post-baseline, 24 months post-baseline
Change in chronic stress as measured by hair cortisol | Baseline, 4-5 months post-baseline, 12 months post-baseline, 24 months post-baseline
Change in psychological violence as measured by Index of Psychological Abuse | Baseline, 4-5 months post-baseline, 12 months post-baseline, 24 months post-baseline

CONTACTS AND LOCATIONS:
Overall Officials: Laura Murray, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Serenity Harm Reduction Programme Zambia (SHARPZ), Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Murray LK, Kane JC, Glass N, Skavenski van Wyk S, Melendez F, Paul R, Kmett Danielson C, Murray SM, Mayeya J, Simenda F, Bolton P. Effectiveness of the Common Elements Treatment Approach (CETA) in reducing intimate partner violence and hazardous alcohol use in Zambia (VATU): A randomized controlled trial. PLoS Med. 2020 Apr 17;17(4):e1003056. doi: 10.1371/journal.pmed.1003056. eCollection 2020 Apr. PMID 32302308